CLINICAL TRIAL: NCT05511974
Title: BASET Scoring: A Novel Simple Biometric Score and Potential Tool for Diagnosis and Grading of Obstructive Sleep Apnea Syndrome Patients
Brief Title: BASET Scoring: A Novel Simple Biometric Score and Potential Tool for Diagnosis and Grading of Obstructive Sleep Apnea Syndrome (OSAS) Patients
Acronym: BASET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amira attia, lecturer of oral and maxillofacial surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R.22.06.1737
Record Dates: First submitted 2022-08-09; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- obstructive sleep apnea patients (Other): Group I : consist of sixty-three patients having OSA. Group II : consist of sixty-three non-OSA patients.
  Interventions: Diagnostic Test: BASET score

INTERVENTIONS:
Diagnostic Test: BASET score — The patients were divided into two groups. Group I (study group): consist of sixty-three patients having OSA. Group II (control group): consist of eighty-one non-OSA patients

SUMMARY:
this study aims to assess the validity of BASET scoring as a new potential tool for diagnosis and grading the severity of OSAS patients and as screening of the risk factors of OSAS.

DETAILED DESCRIPTION:
The study will be conducted on one hundred twenty-six patients attending to sleep disorders breathing Unit, Chest Department at Mansoura University Hospital confirmed by polysomnography

ELIGIBILITY:
Inclusion Criteria:

* All adult patients after having full night polysomnography.

Exclusion Criteria:

* Pregnant patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
assess the performance of BASET score for diagnosis of OSAS | up to 2 weeks.
  assess the performance of BASET score for diagnosis OSAS Region is neither concave nor dark red will take score (0). Region which is dark red but not concave will take score (1). Region which is concave but not dark red will take score (2). Region which is dark red and concave will take score (3).
grading of the severity of OSAS patients. | up to one week
  grading of the severity of OSAS patients. Region is neither concave nor dark red will take score (0). Region which is dark red but not concave will take score (1). Region which is concave but not dark red will take score (2). Region which is dark red and concave will take score (3).

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
The study will be conducted on one hundred twenty-six patients attending to sleep disorders breathing Unit, Chest Department at Mansoura University Hospital confirmed by polysomnography. The patients will be divided into two groups:
  Group I (study group): consist of sixty-three patients having OSA. Group II (control group): consist of sixty-three non-OSA patients.

REFERENCES:
- [Derived] Saleh AM, Ahmed MA, El Said EA, Awadalla NJ, Attia AAMM. BASET scoring: A novel simple biometric score for screening and grading obstructive sleep apnea. Sleep Med X. 2023 Aug 14;6:100083. doi: 10.1016/j.sleepx.2023.100083. eCollection 2023 Dec 15. PMID 37635707